CLINICAL TRIAL: NCT03841292
Title: Using Non-invasive Brain Stimulation (tDCS) to Improve the Effectiveness of Varenicline for Treating Tobacco Dependence: a Randomized Controlled Trial
Brief Title: Using Non-invasive Brain Stimulation (tDCS) With Varenicline for Treating Tobacco Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Laurie Zawertailo, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB #044/2016
Record Dates: First submitted 2019-01-08; First posted 2019-02-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Tobacco Dependence; Smoking Cessation; Tobacco Smoking; Tobacco Use Disorder; Substance Use Disorders; Molecular Mechanisms of Pharmacological Action; Physiological Effects of Drugs
Keywords: Smoking Cessation Medication; Smoking Treatment; Tobacco Treatment; Quitting Smoking; Varenicline; Transcranial Direct Current Stimulation; Neuroimaging; fMRI; Attentional Bias; Eye-tracking; Dependence; Addiction; Cigarettes; Biochemical Confirmation; Cue reactivity; Reward Anticipation; Diffusion Tensor Imaging; Resting State Functional Connectivity; BOLD fMRI; Quantitative T1
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Tobacco Smoking; Substance-Related Disorders; Behavior, Addictive | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: Sham Controlled Randomized Trial
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS+Varenicline (Active Comparator): Active 2mA tDCS (Nuraleve, Canada) with the anode placed over the left dorsolateral prefrontal cortex (dlPFC) and the cathode placed over the right dlPFC for 20 minutes per session. Daily stimulation between Monday to Friday for the first two weeks and then booster sessions every other week for the next 10 weeks.
  Interventions: Drug: Varenicline; Device: Active tDCS
- Sham tDCS+Varenicline (Sham Comparator): Sham tDCS (Nuraleve, Canada)(30 seconds of 2mA and 19.5 minutes of 0 mA) with the anode placed over the left dorsolateral prefrontal cortex (dlPFC) and the cathode placed over the right dlPFC for 20 minutes per session. Daily stimulation between Monday to Friday for the first two weeks and then booster sessions every other week for the next 10 weeks.
  Interventions: Drug: Varenicline; Device: Sham tDCS

INTERVENTIONS:
Drug: Varenicline — Varenicline (Champix®), Pfizer Canada Inc., Kirkland, Quebec. Dispense for 12 weeks. One tablet (0.5mg) once daily for first three days, then one tablet (0.5 mg) twice daily for next four days, then 1 mg (one 1mg tablet) twice daily for the remainder of 12 weeks. Dose adjustments due to adverse events will be allowed (i.e. decrease to 0.5 mg twice daily).
  Other Names: Champix
Device: Active tDCS — Active 2mA tDCS (Nuraleve, Canada) with the anode placed over the left dorsolateral prefrontal cortex (dlPFC) and the cathode placed over the right dlPFC for 20 minutes per session
  Arms: Active tDCS+Varenicline
Device: Sham tDCS — Shame tDCS (Nuraleve, Canada) (30 seconds of 2mA and 19.5 minutes of 0 mA) with the anode placed over the left dorsolateral prefrontal cortex (dlPFC) and the cathode placed over the right dlPFC for 20 minutes per session.
  Arms: Sham tDCS+Varenicline

SUMMARY:
The addition of tDCS as an adjunct to pharmacotherapy is a novel approach but one that is grounded in a growing evidence-base.The primary objective of this research is to provide preliminary evidence of the effectiveness of tDCS as an adjunct treatment to pharmacotherapy for smoking cessation. The investigators hypothesize that the addition of active tDCS to the left DLPFC will improve the effectiveness of varenicline as reflected by higher quit rates at end of treatment compared to the sham group. Smoking status will be biochemically confirmed at various time points using expired cotinine measures. Furthermore, the investigators will be collecting neuroimaging (fMRI) data as well as measures of attentional bias to explore the neurological and physiological correlates from using adjunct tDCS and varenicline therapy.

DETAILED DESCRIPTION:
While varenicline on its own is the most effective medication for smoking cessation, long-term abstinence is still relatively poor. The primary objective of this study is to evaluate the effectiveness of adjunct active tDCS with varenicline in treating tobacco dependence. This study is a double-blind, sham-controlled, randomized clinical trial where 50 daily dependent treatment seeking smokers will be recruited at the Nicotine Dependence Clinic in Toronto, Canada. Participants will be receiving twelve weeks of varenicline treatment (1mg b.i.d.) and randomized 1:1 to either active tDCS (active: 20 minutes at 2 mA) or sham tDCS (30 seconds at 2 mA, 19.5 minutes at 0 mA), daily (M-F) for the first 2 weeks and then every 2 weeks for the next 10 weeks. There will be 2 fMRI scans at baseline and 1 scan at end-of-treatment. Eye-tracking viewing tests will be conducted at baseline, weeks 4, 8, 12 and at 6 months follow up. During the 6 month follow-up, participants will be answering questions regarding their smoking behaviour and craving. Smoking status will be biochemically confirmed at each study visit using expired cotinine.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Aged 19-65
* Treatment seeking smoker
* Daily smoker of CPD>8
* Able to attend daily appointments for tDCS for the first 2 weeks and booster sessions for the next 10 weeks.
* Wiling to undergo 3 fMRI sessions

Exclusion Criteria:

* Current/recent DSM-IV Axis I diagnosis
* Current use of psychoactive drugs or medications
* History of seizures/epilepsy
* Current use of NRT, e-cigarettes or other medications for smoking cessation
* Metal embedded in skull or implanted electrical devices
* No head injury (concussion or loss of consciousness for more than an hour)
* Contraindications to fMRI
* Contraindications to varenicline

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in smoking status over time | At weeks 12 and 26 following start of treatment
  30 Day Continuous abstinence confirmed by expired CO </= 4 ppm

SECONDARY OUTCOMES:
Change in functional brain activation during cognitive tasks | At baseline and 12 weeks following start of treatment
  change in fMRI BOLD response in the brain in response to smoking cues or when anticipating a monetary reward
Change in preference of attention towards visual cues | At weeks 4,8, 12 and 26 weeks following start of treatment.
  Attentional bias to smoking cues, negative/positive cues and high-risk cues measured using an automated eye-tracking apparatus

OTHER OUTCOMES:
Change in brain neurocircuitry over time | At baseline and 12 weeks following start of treatment
  Differences in water diffusion in the brain when participants are at rest in a MRI scanner.
Change in dynamic functional connectivity of the brain at rest over time | At baseline and 12 weeks following start of treatment
  Related to differences in resting state functional brain networks when participants are not doing an explicit task in a fMRI scanner.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A Zawertailo, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Zawertailo L, Zhang H, Rahmani N, Rajji TK, Selby P. Active versus sham transcranial direct current stimulation (tDCS) as an adjunct to varenicline treatment for smoking cessation: Study protocol for a double-blind single dummy randomized controlled trial. PLoS One. 2022 Dec 8;17(12):e0277408. doi: 10.1371/journal.pone.0277408. eCollection 2022. PMID 36480510